CLINICAL TRIAL: NCT05965375
Title: Risk Stratification Value of Biomarkers in Patients With Ventricular Arrhythmias (FUTURE): an Investigator-initiated, National, Multicenter, Retrospective-prospective, Cohort Study
Brief Title: Risk Stratification Value of Biomarkers in Patients With Ventricular Arrhythmias
Acronym: FUTURE
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: 521 Hospital of NORINCO Group (Other); Shaanxi Provincial People's Hospital (Other); Xiangyang Central Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-171
Record Dates: First submitted 2023-07-06; First posted 2023-07-28 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Arrythmia
Keywords: Ventricular Arrhythmia; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, feces and urine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Occasional premature ventricular contractions group: Premature ventricular contractions (PVCs) occur when an electrical impulse originates from an ectopic focus within the ventricle or the interventricular septum, causing premature depolarization of the ventricle before the impulse from the sinoatrial node has reached the ventricle. Occasional PVCs refer to PVCs that occur less than 6 times per minute.
  Interventions: Other: Observational; No Interventions were given.
- Frequent premature ventricular contractions group: Premature ventricular contractions (PVCs) occur when an electrical impulse originates from an ectopic focus within the ventricle or the interventricular septum, causing premature depolarization of the ventricle before the impulse from the sinoatrial node has reached the ventricle. Frequent PVCs refer to PVCs that occur more than 6 times per minute.
  Interventions: Other: Observational; No Interventions were given.
- Short runs of ventricular tachycardia group: Premature ventricular contractions (PVCs) occur when an electrical impulse originates from an ectopic focus within the ventricle or the interventricular septum, causing premature depolarization of the ventricle before the impulse from the sinoatrial node has reached the ventricle. Short runs of ventricular tachycardia refer to three or more consecutive PVCs that occur within 30 seconds.
  Interventions: Other: Observational; No Interventions were given.
- Sustained ventricular tachycardia group: Sustained ventricular tachycardia (VT) is defined as ventricular arrhythmia that lasts for at least 30 seconds and has a heart rate exceeding 100 bpm, or requires termination before 30 seconds due to hemodynamic instability.
  Interventions: Other: Observational; No Interventions were given.
- Ventricular fibrillation group: Ventricular fibrillation refers to the complete disappearance of QRS waves, ST segments, and T waves in the ECG, replaced by different shapes, varying amplitudes, and extremely irregular ventricular fibrillation waves.
  Interventions: Other: Observational; No Interventions were given.

INTERVENTIONS:
Other: Observational; No Interventions were given. — Observational; No Interventions were given.

SUMMARY:
The investigation of biomarkers for immune status and metabolic state, as well as host microbiota composition, in patients with ventricular arrhythmias before and after radiofrequency ablation, can provide new insights for specific and personalized treatment. This can help establish early prediction and prognosis models and provide a basis for clinically effective diagnosis and treatment.

DETAILED DESCRIPTION:
Abnormal immune and metabolic states can lead to the occurrence of various systemic diseases, including the development of cardiovascular diseases through multiple mechanisms. On the other hand, various diseases can also feedback and regulate the immune and metabolic systems. However, currently there is no research on the impact of immune and metabolic states on ventricular arrhythmia. Exploring the biomarker characteristics and risk stratification of patients with ventricular arrhythmias undergoing radiofrequency ablation before and after the procedure can provide new insights for specific and personalized treatment. It can establish early prediction and prognostic models, providing evidence for clinically effective diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ventricular premature beats, ventricular tachycardia, or ventricular fibrillation detected by regular surface twelve-lead electrocardiogram or Holter.

Exclusion Criteria:

* Age <18 or >80 years old;
* Patients with autoimmune diseases or immune deficiencies, or those who have used immunosuppressive or immune modulating agents in the past 3 months;
* Platelet count <100×10^9/L or functional platelet defects;
* Congenital or acquired coagulation or bleeding disorders;
* Patients with a history of organ transplantation or are preparing to receive organ transplantation;
* Unwilling to sign an informed consent or cooperate with the examination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ventricular premature beats, ventricular tachycardia, or ventricular fibrillation detected by regular surface twelve-lead electrocardiogram or Holter.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of MACCE | 3,6 months,1,3,5 years after enrollment.
  Major adverse cardiovascular and cerebrovascular events, including myocardial infarction, stroke, vessel revascularization and all-cause death. The MACCE will be assessed from the medical records.

SECONDARY OUTCOMES:
Change in the incidence of myocardial infarction | 3,6 months,1,3,5 years after enrollment.
  Myocardial infarction diagnosed by clinical doctors will be assessed from the medical records.
Change in the incidence of stroke | 3,6 months,1,3,5 years after enrollment.
  Stroke diagnosed by clinical doctors will be assessed from the medical records.
Change in the incidence of vessel revascularization | 3,6 months,1,3,5 years after enrollment.
  Vessel revascularization assessed by clinical doctors will be assessed from the medical records.
Change in the incidence of all-cause death | 3,6 months,1,3,5 years after enrollment.
  All-cause death diagnosed by clinical doctors will be assessed from the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Chaofeng Sun, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China